CLINICAL TRIAL: NCT01214863
Title: Clinical Results With the AcrySof Toric Intraocular Lens (IOL)
Brief Title: AcrySof Toric Clinical Results
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: M07-007
Record Dates: First submitted 2008-08-07; First posted 2010-10-05 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2010-10

CONDITIONS: Cataracts; Astigmatism
Keywords: Toric Intraocular Lens (IOL)
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- T3: Model SN60T3 assigned by AcrySof Toric calculator
  Interventions: Device: T3
- T4: Model SN60T4 assigned by AcrySof Toric calculator
  Interventions: Device: T4
- T5: Model SN60T5 assigned by AcrySof Toric calculator
  Interventions: Device: T5

INTERVENTIONS:
Device: T3 — Implantation of the AcrySof Toric Intraocular Lens (IOL) Model SN60T3
  Groups: T3
Device: T4 — Implantation of the AcrySof Toric Intraocular Lens (IOL) Model SN60T4
  Groups: T4
Device: T5 — Implantation of the AcrySof Toric Intraocular Lens (IOL) Model SN60T5
  Groups: T5

SUMMARY:
This study is an evaluation of visual outcomes of subjects implanted with the AcrySof Toric Intraocular Lenses (IOLs) Models SN60T3, SN60T4, and SN60T5.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cataracts; has astigmatism falling in range of AcrySof Toric lens as assessed by the AcrySof Toric calculator

Exclusion Criteria:

* Ocular comorbidities affecting visual outcome data,
* Prior refractive surgery,
* Irregular astigmatism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population chosen from physician's patients implanted with the AcrySof Toric intraocular lens (IOL)
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1 day to 6 months

SECONDARY OUTCOMES:
Postoperative refractive cylinder | 1day to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Holladay JT, Wilcox RR, Koch DD, Wang L. Astigmatism analysis and reporting of surgically induced astigmatism and prediction error. J Cataract Refract Surg. 2022 Jul 1;48(7):799-812. doi: 10.1097/j.jcrs.0000000000000871. PMID 35749069